CLINICAL TRIAL: NCT03316664
Title: Assessment of Efficacy of a Psychological Therapy in Inpatients With a Schizophrenic Psychosis
Acronym: CBTSZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Stephan T. Egger, MD, Psychiatric University Hospital, Zurich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBTSZ
Record Dates: First submitted 2017-10-02; First posted 2017-10-20 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychotic Disorders
Keywords: cognitive behavioural therapy; psychotic disorder; schizophrenia; schizoaffective disorder; psychological intervention
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: An 8-week, randomized, controlled, assessor-blind, three-parallel-arm trial is planned with patients diagnosed with a schizophrenic psychosis.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- INT (Experimental): Integrated Neurocognitive Therapy (INT) is a manualized psychological intervention that consists of 30 sessions administered by a therapist and a co-therapist in an open group of 6-8 patients. Sessions will take place twice a week, and each session should last 90 min.
  Interventions: Behavioral: Integrated Neurocognitive Therapy (INT)
- IPT (Active Comparator): Integrated Psychological Therapy (IPT) is a manualized psychological intervention that consists of 5 modules which can be completed in a variable number of sessions that will be administered by a therapist and a co-therapist in an open group of 6- 8 patients. Sessions will take place twice a week, and each session should last 60 to 90 min.
  Interventions: Behavioral: Integrated Psychological Therapy (IPT)
- CoC (Other): COGPACK is a computer-based neuropsychological cognitive training program. It will be administered by a trainer in an open group of 6- 8 patients. Sessions will take place twice a week, and each session will last 45 - 60 minutes.
  Interventions: Other: COGPACK

INTERVENTIONS:
Behavioral: Integrated Neurocognitive Therapy (INT) — Information already included in arm/group description.
  Arms: INT
Behavioral: Integrated Psychological Therapy (IPT) — Information already included in arm/group description.
  Arms: IPT
Other: COGPACK — Information already included in arm/group description.
  Arms: CoC

SUMMARY:
This randomised three-arm study aims to evaluate the efficacy and feasibility of a cognitive behavioral therapy (INT-Integrated Neurocognitive Therapy for Schizophrenia Patients) in the treatment of schizophrenia patients in an inpatient setting. The intervention will be compared with an active comparator (IPT- Integrated Psychological Therapy) and a control condition. Overall the study will include 90 patients (30 in each arm). Each patient will receive at least 16 sessions of the respective treatment. Baseline and follow up assessments up to 12 months after the intervention will investigate the stability of treatment.

DETAILED DESCRIPTION:
Psychotic disorders, and particularly schizophrenia, are severe psychiatric disorders, characterized by psychotic symptoms (mainly hallucinations and delusions), disorganized speech, thought and behavior, and negative symptoms like blunted affect. People who have schizophrenia are chronically impaired. Schizophrenia is one of the first causes of disability worldwide with enormous direct and indirect costs.

The introduction of antipsychotics revolutionized the treatment and care of schizophrenia patients; remaining the cornerstone of schizophrenia treatment. Although new antipsychotics were introduced, they share the same mechanism of action (dopamine D2 antagonism). To date, nearly one-third to half of the patients still do not or respond poorly to antipsychotic treatment; furthermore, some core symptoms of the disorder are not fully addressed by this type of medication.

Parallel to pharmacological treatments, there has been a steady research in psychological interventions for schizophrenia. Current interventions had a more biologic understanding of the disorder and adopted a diathesis-stress model to explain symptoms and course, incorporating adaptation and adjustment through learned and practiced coping strategies. There are many psychological treatments for schizophrenia, although all are considered roughly equivalent, empirical data shows slight differences in efficacy; in particular, Cognitive Behavioural Therapy (CBT) yields small to medium sized effects in addition to psychopharmacological treatment.

There are several available manualized psychological group interventions for patients with a schizophrenic psychosis. One the is the "Integrated Psychological Therapy for Schizophrenia Patients (IPT)", it was developed and introduced into clinical practice almost 30 years ago. It combines neurocognitive and social cognitive interventions with social skills and problem- solving approaches, it has been extensively evaluated by several independent groups, in inpatient and outpatient settings as well, showing an overall improvement in participants.

During the last decade, the cognitive section of IPT was further developed, with the "Integrated Neurocognitive Therapy for schizophrenia patients (INT)" was the final result of this process, with the peculiarity that it was designed to fit the needs of outpatients. While IPT focuses predominantly on the domains of speed of processing, attention, reasoning, and problem-solving as well as on emotion and social perception; INT in contrast targets all 11 neuro- and social-cognitive MATRICS-domains. Furthermore, INT uses computerized neurocognitive exercises for restitution. Initial trials seem to confirm INT as a feasible and efficient group therapy approach with the potential to improve functional outcome in schizophrenia outpatients

The investigators, plan investigational trial to assess the efficacy and feasibility of INT for patients with schizophrenia in an inpatient setting. Therefore, an 8-week, randomized, controlled, assessor-blind, three-parallel-arm trial is planned with patients diagnosed with a schizophrenic psychosis. Following baseline assessment, patients will be randomly assigned to either IPT, INT or a control intervention.

All study interventions, i.e.: the experimental intervention, the psychological control intervention, and the control condition will occur simultaneously twice a week to avoid participants from involuntarily switch groups. Therapists of the psychological experimental and control intervention, as well as trainers involved in the control condition, are not involved in the recruitment, assessment, and assignment of participants of the study. Study interventions will be held in group sessions with 6 to 8 participants each; we plan to conduct five such batches till we reach our sample size of at least 30 participants in each intervention arm.

Patients undergoing psychological interventions should have some prerequisites and conditions which make them suitable for the intervention; this, however, is not fully compatible with a random allocation of participants. Through randomization there is the possibility that participants are not able to cope with their assigned treatment; therefore in a pragmatic way patients will be allowed to switch in another treatment arm. Accordingly after two weeks; patients will be reassessed; reallocation will be followed according to predefined criteria for excessive demands or under requirement.

Participants which switch groups should complete the 8-week intervention in the second assigned group. The assessment at week two will be considered their baseline, with subsequent measures eight weeks later analog to those who did not switch treatment groups. For the final analysis and to preserve randomization the data from those who did not switch treatment groups will be analyzed: however data from the switching groups will be analyzed separately in an ITT fashion.

ELIGIBILITY:
Inclusion Criteria:

* Participants are competent to give informed consent.
* Diagnosis of Schizophrenia or Schizoaffective Disorder (ICD-10).
* Participants are between 18 and 65 years of age.
* Fulfillment of regular compulsory education.
* German language proficiency as a native speaker or level B1

Exclusion Criteria:

* Unwilling or unable to comply with study instructions.
* Low Intelligence as stated by failure to accomplish regular compulsory education.
* Currently in another psychotherapeutic treatment, either in individual or group sessions.
* Current consumption of Alcohol or illicit Drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Symptomatology at 12 Months. | Baseline, 2 Weeks, 10 Weeks, 6 Months, and 12 Months.
  The "Positive and Negative Syndrome Scale" (PANSS) was designed to measure the severity of psychopathology in adult patients with a psychotic disorder, mainly schizophrenia and schizoaffective disorder.

SECONDARY OUTCOMES:
Change from Baseline Symptomatology at 12 Months. | Baseline, 2 Weeks, 10 Weeks, 6 Months, and 12 Months.
  The Mini-ICF (mICF) was developed to classify disorders according to the level of functioning and capacity in an abbreviated version.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Redlich Bossy M, Mueller D, Seifritz E, Vetter S, Egger ST. Feasibility and Efficacy of a Psychological Therapy for Patients With a Schizophrenic Psychosis in an Inpatient Setting: Study Protocol of a Randomized Switch Controlled Trial. Front Public Health. 2020 Aug 12;8:391. doi: 10.3389/fpubh.2020.00391. eCollection 2020. PMID 32903368